CLINICAL TRIAL: NCT06059625
Title: RECURRENCE OF ROTATOR CUFF LESION AFTER SURGICAL REPAIR WITH SINGLE-ROW vs DOUBLE-ROW SUTURE BRIDGE TECNIQUE: A COMPARATIVE STUDY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CUFFIA3T
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Cuff Injury, Rotator
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DOUBLE-ROW (Experimental): rotatori cuff repair with double-row suture bridge technique
  Interventions: Procedure: rotatori cuff repair
- SINGLE-ROW (Active Comparator): rotatori cuff repair with single-row technique
  Interventions: Procedure: rotatori cuff repair

INTERVENTIONS:
Procedure: rotatori cuff repair — rotatori cuff repair

SUMMARY:
The rotator cuff is a muscle-tendon complex consisting of the tendons of the supraspinatus, subspinatus, subscapularis, and small round muscles capable of allowing movement of the shoulder joint in the various planes of space and stabilizing the glenohumeral joint.

Rotator cuff tendon injuries are very common. In most cases, these injuries are mostly degenerative based, as they are related to the aging process of the individual. However, it is increasingly common to diagnose such injuries in young individuals as well.

The reported incidence of rotator cuff injuries ranges from 5% to 40%, and of course the prevalence increases with age until it reaches 51% in patients older than 80 years.

The diagnosis of rotator cuff injury is made based on clinical examination and instrumental investigations such as Nuclear Magnetic Resonance Imaging (MRI).

Rotator cuff repair involves the use of anchors with included suture threads that allow the tendons to be returned to the level of the anatomical insertion, called the footprint.

Suture technique varies depending on the extent of injury and tendon and bone quality.

Single-row (single row) or double-row suture bridge (double-row suture bridge) anchoring techniques are currently a hotly debated topic in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥45 years with a diagnosis of full-thickness rotator cuff injury <2cm
* Arthroscopic rotator cuff repair surgery with single row or double row suture bridge
* Follow-up > 24 months
* Completeness of clinical-radiographic documentation
* Patients at first rotator cuff repair surgery on affected side

Exclusion Criteria:

* Patients with associated injuries to the affected upper limb
* Patients with neuromuscular disorders, or established psychomotor disorders
* Patients with associated injuries of the subscapularis muscle tendon
* Patients with a history of previous surgery of the affected shoulder
* Patients with massive rotator cuff injury > 2cm
* Patients with severe pathologies of other organs or apparatuses that limit competitive or recreational sports activities
* Pregnant women
* Patients who cannot undergo high-field MRI (pcs with cochlear implants, cardiac, vascular or osteoarticular magnetic, pcs with previous gunshot wounds)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
radiological outcome (Sugaya score) | 24 months
  The Sugaya classification is used to evaluate rotator cuff repair, assessing post-operative rotator cuff repair on oblique coronal, oblique sagittal and transverse MRI planes.
  Scores range from 0 to 5 with a score of 0 indicating better tendon quality and no lesion and 5 indicating worse tendon quality with complete lesion.
clinical outcome (American Shoulder and Elbow Surgeons shoulder score) | 24 months
  ASES score is designed to assess the condition of the shoulder, regardless of disease pathology, requiring both a physician assessment and a patient-completed portion.
  Scores range from 0 to 100 with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition.
clinical outcome (University of California and Los Angeles shoulder score) | 24 months
  UCLA shoulder score is a jointly completed score, with both physician and patient completed portions.
  Scores range from 0 to 35 with a score of 0 indicating worse shoulder function and 35 indicating better shoulder function.
clinical outcome (Costant-Murley score) | 24 months
  The Costant-Murley score is designed to assess the functional state of a normal, a diseased, or a treated shoulder. It contains both physician-completed and patient-reported portions.
  Scores range from 0 points (most disability) to 100 points (least disability).
clinical outcome (Range Of Motion) | 24 months
  ROM expresses in degrees the degree of range of motion that a joint can perform along its full range of motion whether active or passive through an external aid.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Khoriati AA, Antonios T, Gulihar A, Singh B. Single Vs Double row repair in rotator cuff tears - A review and analysis of current evidence. J Clin Orthop Trauma. 2019 Mar-Apr;10(2):236-240. doi: 10.1016/j.jcot.2019.01.027. Epub 2019 Jan 30. No abstract available. PMID 30828184
- [Result] Padua R, Padua L, Ceccarelli E, Bondi R, Alviti F, Castagna A. Italian version of ASES questionnaire for shoulder assessment: cross-cultural adaptation and validation. Musculoskelet Surg. 2010 May;94 Suppl 1:S85-90. doi: 10.1007/s12306-010-0064-9. PMID 20383686
- [Result] Sugaya H, Maeda K, Matsuki K, Moriishi J. Functional and structural outcome after arthroscopic full-thickness rotator cuff repair: single-row versus dual-row fixation. Arthroscopy. 2005 Nov;21(11):1307-16. doi: 10.1016/j.arthro.2005.08.011. PMID 16325080